CLINICAL TRIAL: NCT02994342
Title: Efficacy, Tolerability and Safety of a New Medical Device, Zp-025 Vaginal Gel, in the Treatment of Vaginal Dryness in Post-menopausal Women With Vaginal Atrophy
Brief Title: Efficacy and Tolerability Study of ZP-025 Vaginal Gel for the Treatment of Vaginal Dryness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z7213M02
Record Dates: First submitted 2016-12-01; First posted 2016-12-15 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Vaginal Dryness
Keywords: vaginal dryness; vaginal gel; colostrum; vaginal atrophy
MeSH Terms: interventions — Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal gel, Medical Device Class 2A (Active Comparator): Every subject has been treated for 56 consecutive days, twice daily with a vaginal application
  Interventions: Device: Vaginal gel, Medical Device Class 2A
- Lifestyle counseling (No Intervention): Every subject has been observed for 56 consecutive days

INTERVENTIONS:
Device: Vaginal gel, Medical Device Class 2A — Application twice a day of vaginal gel for 56 consecutive days
  Other Names: Monurelle Biogel
  Arms: Vaginal gel, Medical Device Class 2A

SUMMARY:
Evaluation of ZP-025 vaginal gel in terms of efficacy and safety in the treatment of vaginal dryness in post-menopausal women with vaginal atrophy in comparison to a group of non-treated post-menopausal women with vaginal atrophy after 56 consecutive days and at 4-week follow-up only for women applying ZP-025 vaginal gel.

DETAILED DESCRIPTION:
Evaluation of ZP-025 vaginal gel in terms of efficacy, tolerability and safety in the treatment of vaginal dryness in post-menopausal women with vaginal atrophy in comparison to a group of non-treated post-menopausal women with vaginal atrophy for 56 consecutive days.

This trial will be conducted in compliance with last version of Declaration of Helsinki, with GCP as applicable to investigations with IMD, with the applicable regulatory requirements and with CRO and Sponsor's SOPs.

This is a multi-centre, national, randomized, controlled vs. no-treatment, open label study The study will take place in 6 centers of menopause at public Hospitals/Universities. An ancillary study will be carried on for subjects randomized to ZP-025 group with a follow-up visit at 4 weeks

ELIGIBILITY:
Inclusion Criteria:

* caucasian women <70 years, in physiological postmenopausal status for at least 2 years;
* women with signs and symptoms of vaginal atrophy (i. e. vaginal discomfort, itching, dyspareunia, dryness);
* signed informed consent; willing and able to comply with study procedures

Exclusion Criteria:

* childbearing potential women;
* ascertained or presumptive hypersensitivity to the formulation ingredients;
* therapy with systemic or vaginal oestrogens within 6 months from the inclusion;
* current urinary or vaginal infection (cultural positive result to vaginal or urines microbiological swab in the 7 days preceding inclusion);
* previous episodes of vaginal bleeding or spotting in the last 6 months;
* vaginal prolapse and any other disease that could interfere with the study conduction and participation

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in subjective symptoms of total score related to vaginal discomfort | 56 days
  Change in subjective symptoms of total score related to vaginal discomfort (vaginal dryness, vaginal and/or vulvar irritation/itching, vaginal soreness, dysuria, and dyspareunia and vaginal bleeding associated with sexual activity) has been recorded on daily diary by subject from baseline to day 56, evaluated using a subjective evaluation scale (VRS at four items: 0= absent, 1= mild, 2=moderate, 3=severe). Each item is summed up to get to a total symptoms score.

SECONDARY OUTCOMES:
change of vaginal health index | 56 days
  change of vaginal health index calculated on the basis of vaginal moistness, vaginal fluid volume, vaginal elasticity, vaginal mucosa, and vaginal pH on a scale ranging from 1 (poorest) to 5 (best) from baseline (day 0), to day 56 recorded by investigator
change of maturation index | 56 days
  change of maturation index: parabasal, intermediate and superficial cells from baseline (day 0) to day 56
change of Female Sexual Function Index | 56 days
  change of Female Sexual Function Index (FSFI) from baseline to day 56 in women with at least one sexual intercourse in the treatment period recorded by subject
change in each subjective symptom score related to vaginal discomfort | 56 days
  change in each symptom score from baseline to end of study recorded on daily diary by subject(vaginal dryness, vaginal and/or vulvar irritation/itching, vaginal soreness, dysuria, and dyspareunia and vaginal bleeding associated with sexual activity) has been recorded on daily diary by subject from baseline to day 56, evaluated using a subjective evaluation scale (VRS at four items: 0= absent, 1= mild, 2=moderate, 3=severe).
local tolerability and incidence of adverse events | 56 days
  local tolerability registered daily by subject in the subject's diary during the application; period and by the investigator from baseline to day 56; AEs registered over all study period (first patient in - last patient out) - In particular the following assessments will be done: vital signs during all visits. transvaginal ecography to exclude any possible endometrial disease or endometrial thickness variation at the screening visit and at the end of the study, clinical evaluation by the investigator at all visits.
change of Female Sexual Distress Scale-Revised | 56 days
  change of Female Sexual Distress Scale-Revised (FSDS-R revised 2005) from baseline (Day 0) to day 28 and to the end of the study in women with at least one sexual intercourse in the treatment period recorded by subject
change of cariopicnotic index (CPI), | 56 days
  change of cariopicnotic index (CPI), as a correlation of superficial cells with picnotic nuclear and general amount of cells ratio, expressed in percentage from baseline (day 0), to day 56

CONTACTS AND LOCATIONS:
Overall Officials: Rossella Nappi, Md PhD, Study Director — Obstetrics and Gynaecology Clinic IRCCS Fondazione San Matteo University of Pavia, Italy
Locations (6):
- Italy (6):
  - Ospedale San Giovanni di Dio, Cagliari
  - Policlinico Careggi, Florence
  - Clinica Macedonio Melloni, Milan
  - Policlinico di Modena, Modena
  - Policlinico Federico II, Napoli
  - Policlinico San Matteo, Pavia

IPD SHARING:
Plan to Share IPD: Yes
IPD should be requested to sposnor contacts

REFERENCES:
- [Derived] Nappi RE, Cagnacci A, Becorpi AM, Nappi C, Paoletti AM, Busacca M, Martella S, Bellafronte M, Tredici Z, Di Carlo C, Corda V, Vignali M, Bagolan M, Sardina M. Monurelle Biogel(R) vaginal gel in the treatment of vaginal dryness in postmenopausal women. Climacteric. 2017 Oct;20(5):467-475. doi: 10.1080/13697137.2017.1335703. Epub 2017 Jun 28. PMID 28657769